CLINICAL TRIAL: NCT02725970
Title: Healthy Eating and Lifestyle for Total Health
Acronym: HEALTH
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Theresa A Nicklas, Professor of Pediatrics, Baylor College of Medicine
Other Study IDs: H-23839
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Eating Behavior
Keywords: HEALTH; barriers; facilitators; DGA; BMI; Public Schools
MeSH Terms: conditions — Feeding Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Children's Nutrition Research Center: Survey, no intervention.
  Interventions: Other: survey
- Western Human Nutrition Research Center: Survey, no intervention.
  Interventions: Other: survey
- Human Nutrition Research Center On Aging: Survey, no intervention.
  Interventions: Other: survey
- Delta Obesity Prevention Research Center: Survey, no intervention.
  Interventions: Other: survey
- Beltsville Human Nutr Research Center: Survey, no intervention.
  Interventions: Other: survey
- Grand Forks Human Nutr Research Center: Survey, no intervention.
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — Cross-sectional survey

SUMMARY:
The Dietary Guidelines for Americans provide recommendations for making better food and physical activity choices that promote health and help prevent disease. Yet, few Americans meet the Dietary Guidelines for Americans (DGA) and a large percentage are overweight.

DETAILED DESCRIPTION:
The goal of the research was to examine the association between weight and the barriers and facilitators to meeting the DGA in a multi-site study using a cross-sectional survey. 836 caregiver-child dyads enrolled and completed the HEALTH study questionnaire across six sites among three race/ethnic groups participating in the HEALTH Study. Barriers and facilitators to meeting the DGA were assessed using a validated questionnaire which was developed specifically for the HEALTH Study. Heights and weights were measured. A series of bivariate regression analyses were conducted to examine the association between the caregivers BMI or the children BMI z-score and the barriers and facilitators to meeting the DGA, adjusting for appropriate covariates in the models. Path analysis was used to examine the relationship of caregivers and children barriers and facilitators to their relative BMI.

ELIGIBILITY:
1. Children in grade 5 and primary caregiver of a child in the 5th grade (the primary caregiver was defined as the person responsible for the health of the child and who has the most influence in what the child eats most days of the week)
2. Attend public school and caregiver to a child in a public school
3. Fell in one of three racial/ethnic groups (African Americans, Hispanics, White)

Exclusion Criteria:

1. Pregnant women were not recruited as their dietary intake was different because of pregnancy.
2. Children not attending 5th grade in public school.
3. Parents of children not attending 5th grade in public school
4. parents of children attending 5th grade in public school but who were not responsible for the health of the child and who did not have the most influence in what the qualified child ate most days of the week.

Ages: 8 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Fifth-grade children and their caregivers, or a caregiver of a 5th grade child attending a public school.
Sampling Method: Non-Probability Sample
Enrollment: 836 (Actual)
Dates: Start 2011-01; Primary Completion 2012-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Measuring and Reporting on the Barriers and Facilitators to Meeting the Dietary Guidelines of Americans among 5th Graders and the Caregivers of 5th Graders Was Assessed Using Questionnaires. | 3/2010- 7/2012

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Nicklas, DrPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- USDA/ARS Children's Nutrition Research Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicklas TA, Jahns L, Bogle ML, Chester DN, Giovanni M, Klurfeld DM, Laugero K, Liu Y, Lopez S, Tucker KL. Barriers and facilitators for consumer adherence to the dietary guidelines for Americans: the HEALTH study. J Acad Nutr Diet. 2013 Oct;113(10):1317-31. doi: 10.1016/j.jand.2013.05.004. Epub 2013 Jul 17. PMID 23871110
- [Derived] Nicklas T, Liu Y, Giovanni M, Jahns L, Tucker K, Laugero K, Bogle M, Chester D. Association between barriers and facilitators to meeting the Dietary Guidelines for Americans and body weight status of caregiver-child dyads: the Healthy Eating and Lifestyle for Total Health Study. Am J Clin Nutr. 2016 Jul;104(1):143-54. doi: 10.3945/ajcn.115.123372. Epub 2016 May 18. PMID 27194306